CLINICAL TRIAL: NCT00103571
Title: Olanzapine Versus Aripiprazole in the Treatment of Acutely Ill Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8928; F1D-US-HGLS
Record Dates: First submitted 2005-02-10; First posted 2005-02-11 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Aripiprazole

INTERVENTIONS:
Drug: Olanzapine
Drug: Aripiprazole

SUMMARY:
The purposes of this study are to assess similarities and differences in the efficacy (how well the drug works), safety, and side effects of olanzapine and aripiprazole in patients with schizophrenia, schizoaffective disorder, or schizophreniform disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have schizophrenia, schizoaffective disorder, or schizophreniform disorder
* Patients must be agitated
* Patients must display psychotic symptoms
* Patients must be inpatients who are expected to stay in the hospital for at least 5 days
* Patients must be 18 to 55 years of age

Exclusion Criteria:

* Patients may not be hospitalized for greater than 72 hours prior to study start
* Patients may not have received more than one dose of olanzapine or aripiprazole within 72 hours prior to study start
* Patients may not be actively suicidal
* Patients may not be diagnosed with substance-induced psychosis or substance dependence
* Patients may not have acute, serious, or unstable medical conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600
Dates: Start 2004-07; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to test the hypothesis that olanzapine is superior to aripiprazole in the reduction of symptoms of agitation in acutely ill patients with schizophrenia, as measured by mean change in the
Positive and Negative Syndrome Scale Excited Component (PANSS-EC) over 5 days of treatment (4 continuous 24 hr treatment exposures). The null hypothesis of the study is that there is no difference between olanzapine and
aripiprazole in reducing agitation.

SECONDARY OUTCOMES:
The reduction in positive symptoms as measured by the Brief Psychiatric Rating Scale Positive subscale (PBRS Positive);
The reduction of symptoms of agitation as measured by Overt Agitation Severity Scale (OASS);
The proportion of patients responding to treatment and the time to response based on varying levels in the percent reduction of
the PANSS_EC from baseline;
The reduction in overall severity of psychiatric illness as measured by the Clinical Global Impression-Severity Scale (CGI-S);
The intensity of nursing intervention (e.g. seclusion, restraint, special nursing watch), as measured by the Global Assessment
of Nursing Intervention
The proportion of patients using pm lorazepam and the time-course of usage.
The proportion of patients discontinuing from the study due to lack of efficacy or due to adverse events related to worsening
of psychiatric illness.
Patient satisfaction with their medication, as measured by Drug Attitude Inventory (DA1-10).
A sensitivity analysis will be performed on two randomly chosen subsamples of the overall patient population by analyzing the
primary objective respectively.
Additional secondary objectives of the study are to compare the safety of olanzapine versus aripiprazole over the course of 5
days in the treatment of acutely ill patients with schizophrenia as assessed by:
Relative degree of sedation as measured by the Agitation Calmness Evalution Scale (ACES);
Review of spontaneous (unsolicited) treatment emergent adverse events;
Development of extrapyramidal symptoms as assessed by daily Modified Simpson-Angus and Barnes Akathisia scale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Saint Charles, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Memphis, Tennessee
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Rio Piedras, Puerto Rico

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com